CLINICAL TRIAL: NCT01731834
Title: Pain and Stress Assessment in Children Undergoing Respiratory Physical Therapy Techniques
Brief Title: Pain and Stress Assessment in Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Maria Teresa de Mendonça Biasi, Assessment of pain and stress in children undergoing respiratory physiotherapy, Federal University of Uberlandia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11212PSC014; FUUberlandia (Registry Identifier: FUUberlandia)
Record Dates: First submitted 2012-11-18; First posted 2012-11-22 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Acute Respiratory Infections
Keywords: Pain; Stress; Physiotherapy; Children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspiration of secretion (Active Comparator): 10 children are evaluated at rest, during and after aspiration technique secretion
  Interventions: Other: Vibrocompression and aspiration of secretions
- Vibrocompression (Experimental): 10 children will be assessed at rest, during and after the maneuver vibrocompression
  Interventions: Other: Vibrocompression and aspiration of secretions

INTERVENTIONS:
Other: Vibrocompression and aspiration of secretions — The 20 children, study participants will be randomly assigned to different groups, where 10 children will be evaluated during vibrocompression maneuver, and another 10 will be assessed on the aspiration procedure. Randomization will be performed using an opaque envelope for specifying which group selection technique is evaluated.

SUMMARY:
There may be pain and / or stress with vibrocompression. There may be pain and / or stress with the aspiration of secretions.

DETAILED DESCRIPTION:
Randomization to 10 children and 10 vibrocompression for aspiration of secretion.

Fill in the evaluation form. Monitoring Heart Rate and Peripheral O2 Saturation (rest, during and after the technique performed).

Photographic Record (rest, during and after the technique performed). Saliva Collection (rest, 5, 20 and 40 minutes after running technics). Data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Indication of Respiratory Therapy

Fasting for one hour before the moment of collection

Term of Free and Informed Consent Form (ICF) signed by parents or legal guardians

Exclusion Criteria:

* Children in postoperative period acute

Presence of thoracic drain or mediastinal

Children using drugs to sedative or analgesic purpose of deep sedation

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Assess whether there is pain in children when performed randomized technique | two years
  Rate NIPS - Infant Pain Scale

SECONDARY OUTCOMES:
Assess whether there is stress in children during the technical run | two years
  Biochemical analysis of cortisol and salivary amylase

OTHER OUTCOMES:
Correlate the pain and the stress generated. | two yars
  Also assess heart rate, respiratory rate, and oxygen saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Biasi, Third, Principal Investigator — FUUberlândia
Locations (1):
- FUUberlândia, Uberlândia, Minas Gerais, Brazil